CLINICAL TRIAL: NCT03462446
Title: Estimate of Costs Associated With Atrial Fibrillation Treatment With Rivaroxaban Versus Vitamin K Antagonists
Brief Title: Analysis of the Potential Savings of Rivaroxaban Events Versus Vitamin K Antagonists Events
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18231
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; VKA; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group with Rivaroxaban: Patients treated with Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Control group with VKAs: Patients treated with VKAs. This control group will be subsequently divided based on the TTR value in the last 6 months (below 65% and above 65%).
  Interventions: Drug: Vitamin K antagonists (VKAs)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by treating physicians
  Groups: Treatment group with Rivaroxaban
Drug: Vitamin K antagonists (VKAs) — As prescribed by treating physicians. VKAs are Acenocoumarol and Warfarin.
  Groups: Control group with VKAs

SUMMARY:
The main objective of this project is to evaluate savings in direct costs as regards the use of rivaroxaban versus vitamin K antagonists (VKAs) in routine clinical practice using data from three cohorts of patients receiving VKAs or rivaroxaban in Spain, including the time in therapeutic range (TTR) values of the same and the incidence of events in the first year following diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Diagnosis of non-valvular AF (ICD code 427.31)
* Pharmacological treatment with VKAs or rivaroxaban following diagnosis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Selected population will include records registered in electronic databases of patients diagnosed with nonvalvular AF, receiving treatment with VKAs or rivaroxaban for one year.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range (TTR) values in the last 6 months | 6 months
Presence of stroke | 12 months
  Presence of stroke prior and subsequent to treatment
Active substance received | 12 months
  Rivaroxaban or VKAs (Acenocoumarol and Warfarin)

SECONDARY OUTCOMES:
Date of stroke | 12 months
Type of stroke | 12 months
  Type of stroke acccording to patients group: unknown, haemorrhagic or ischaemic.
Duration of treatment (in days) | 12 months
Dose of the prescribed treatment | 12 months
Frequency of the prescribed treatment (in hours) | 12 months

OTHER OUTCOMES:
Date of AF diagnosis | 12 months
Comorbidities | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Granada, Spain